CLINICAL TRIAL: NCT05205746
Title: Phase II Study to Evaluate Immunogenicity and Safety in Subjects With Evidence of Prior Immunity to SARS-CoV-2 of a Single Intramuscular or Intranasal Dose of the Live Recombinant Newcastle Disease Virus Based AVX/COVID-12 Vaccine
Brief Title: Phase II Study of AVX/COVID-12 Vaccine in Subjects With Prior SARS-CoV-2 Immunity Evidence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorio Avi-Mex, S.A. de C.V. (Industry)
Collaborators: National Council of Science and Technology, Mexico (Other); Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: AVX-SARS-CoV-2-VAC-002
Record Dates: First submitted 2022-01-22; First posted 2022-01-25 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: SARS CoV 2 Infection
Keywords: Newcastle Disease Virus; rNDV; COVID-19; SARS-Cov-2 Vaccine; Booster COVID-19 Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Patients will be assigned according to their previous vaccine.
Who Masked: Participant, Investigator
Masking Description: The first sentinel group (6 of each previous vaccine) will be without masked only to the subjects to ensure safety measurement in each group. The randomized double-mask placebo-controlled phase will begin when the safety committee, after evaluating the information from the sentinel group of the first three subjects (by vaccine and by specific route of administration), gives authorization to continue with the recruitment. It will be conducted through a computerized assignment system. Randomization for the double-masking phase of the study will be carried out using a computer assignment system.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Intramuscular (Experimental): 10 8.0 EID 50/dose intramuscular
  Interventions: Biological: Recombinant NDV Vectored Vaccine for SARS-CoV-2
- Intranasal (Experimental): 10 8.0 EID 50/dose intranasal
  Interventions: Biological: Recombinant NDV Vectored Vaccine for SARS-CoV-2
- Intramuscular Placebo (Other): Physiological saline solution of Sodium Chloride at 0.9% Intramuscular After mask opening ChAdOx-1-S[recombinant]) Intramuscular
  Interventions: Biological: Placebo
- Intranasal Placebo (Other): Physiological saline solution of Sodium Chloride at 0.9% Intranasal After mask opening ChAdOx-1-S[recombinant]) Intramuscular
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Recombinant NDV Vectored Vaccine for SARS-CoV-2 — Recombinant Newcastle Disease Virus Vectored Vaccine for SARS-CoV-2
  Arms: Intramuscular; Intranasal
Biological: Placebo — Physiological saline solution of Sodium Chloride at 0.9% After mask opening ChAdOx-1-S[recombinant]) Intramuscular
  Arms: Intramuscular Placebo; Intranasal Placebo

SUMMARY:
This is a Phase II study with single-blinded safety phase followed by double-blinded randomization, placebo-controlled, of administration of a single dose by two different administration routes (intramuscular route or intranasal route), to evaluate immunogenicity and safety of the recombinant SARS-CoV-2 vaccine (AVX/COVID-12 vaccine) based a live Newcastle disease viral vector (rNDV) in 396 healthy subjects with evidence of prior immunity to SARS-CoV-2, followed by a booster response assessment with an intramuscular dose of COVID-19 vaccine (ChAdOx-1 -S[recombinant]) in subjects originally randomized to the placebo arm at several research sites in Mexico City.

DETAILED DESCRIPTION:
General objective:

To demonstrate immunogenicity due to the administration of a single dose of AVX/COVID-12 vaccine at a dose of 108.0 EID50%/dose by the intramuscular or intranasal route in subjects with evidence of prior immunity to SARS-CoV-2.

Primary objectives:

* To demonstrate an increase in the total titers of neutralizing anti-Spike IgG antibodies in serum, as well as an increase in the proportion of peripheral blood T lymphocytes that produce interferon gamma in response to stimulation with Spike protein or peptides derived from Spike protein, 14 days after intramuscular administration of a single dose of AVX/COVID-12 vaccine (108.0 EID50%/dose) compared to the response obtained after administration of placebo.
* To demonstrate an increase in the total titers of neutralizing anti-Spike IgG antibodies in serum, as well as an increase in the proportion of peripheral blood T lymphocytes that produce interferon gamma in response to stimulation with Spike protein or peptides derived from Spike protein, 14 days after intranasal administration of a single dose of AVX/COVID-12 vaccine (108.0 EID50%/dose) compared with the response obtained after administration of placebo.

Secondary objectives:

* To evaluate serum titers of IgG anti-Spike antibodies and neutralizing anti-SARS-CoV-2 antibodies at 0, 14, 42, 90, 180 and 365 days after intramuscular or intranasal administration of the AVX/COVID-12 vaccine.
* To assess the proportion of proliferating cells and cytokine production by peripheral blood T lymphocytes in response to stimulation with Spike protein at 0, 14, 180 and 365 days after intramuscular or intranasal administration of the AVX vaccine/COVID-12.

Safety objective:

To assess the safety of immunization using a single intramuscularly or intranasally administered dose of AVX/COVID-12 vaccine in subjects with prior immunity to SARS-CoV-2.

Exploratory objectives:

• Evaluation of the increase in the immune response according to the previously defined parameters of anti-Spike IgG antibody titers, serum titers of neutralizing anti-SARS-CoV-2 antibodies, the increase in the proportion of T lymphocytes producing Gamma interferon according to two stratification schemes as long as the number of recruited subjects allows it: A) By underlying technology of the vaccines received prior to enrollment in the study. The three groups of technology to be explored are inactivated viruses, adenoviral vectors, and mRNA-based technology.

B) By specific vaccine received prior to enrollment in the study as long as the number of subjects recruited for each vaccine allows it.

• Evaluation of the local response in nasal mucous for subjects who were randomized to receive vaccination by both routes, which consists of: A) The determination and quantification of IgA anti-Spike antibodies in mucus or epithelial scraping samples or in an oral fluid rinse.

* Evaluation of the appearance of anti-N and anti-S antibodies on days -4, 7, 14, 42, 90, 180 and 365 days after intramuscular or intranasal administration of the AVX/COVID-12 vaccine.
* Evaluation of the incidence of confirmed cases of SARS-CoV-2 infection in study subjects starting from vaccination in a systematic way until day 28 post-vaccination and in a targeted way (in case of suspicious symptoms) until the end of the study.
* Evaluation of the increase in the immune response according to the parameters of anti-Spike IgG-type antibody titers, anti-SARS-CoV-2 neutralizing antibody serum titers and an increase in the proportion of interferon gamma-producing T lymphocytes in subjects who are originally randomized to placebo and subsequently receive an intramuscular boost with COVID-19 vaccine ChAdOx-1-S[recombinant]).

Clinical trial hypothesis:

Intramuscular or intranasal administration of the AVX/COVID-12 vaccine at a dose of 108.0 EID50%/dose in subjects with prior immunity to SARS-CoV-2 (induced by vaccination) produces an increase in total serum antibody titers of type IgG anti-Spike and increases the titers of neutralizing anti-SARS-CoV-2 antibodies, and additionally produces an increase in the proportion of interferon gamma-producing T lymphocytes in response to stimulation with the Spike protein or peptides derived from the Spike protein, when these parameters are analyzed 14 days after administration.

Rationale of the use of the product in clinical research:

Non-clinical studies and the phase I clinical trial have demonstrated the safety of the AVX/COVID-12 vaccine in intramuscular as well as intranasal route of administration. The signals of immunogenicity in animal models are clear. The evaluation of the immune response in healthy volunteers during the Phase I clinical study after the administration of the vaccine either intramuscularly or intranasally demonstrated the immunogenicity of the vaccine, which justifies the advance of the vaccine development program.

Clinical trial design:

A mixed with single-blind low safety phase followed by double-blind randomization, placebo-controlled, single-dose intramuscular or intranasal, phase II study, in subjects with evidence of prior immunity to SARS-CoV-2, followed by a booster response assessment phase with an intramuscular dose of COVID-19 vaccine (ChAdOx-1-S[recombinant]) in subjects originall randomized to the placebo arm. .

Description of the single-blind safety phases and the double-blind randomization placebo-controlled phase and the evaluation phase of the response to the booster with the COVID-10 vaccine (ChAdOx-1-S[recombinant]):

For each arm of the study (intramuscular or intranasal):

A) The safety phase consists of the single-blind assignment (subject blinded) to the arm that receives the AVX/COVID-12 vaccine to the first three subjects of each specific vaccine who are recruited to the study in each arm, intramuscular and intranasal, independently. The first three subjects in each arm will be subjected to a strict safety follow-up during the 7 days after the administration of the vaccine. The safety information collected during those seven days will be evaluated by an independent safety committee who will decide if it is necessary to stop the study of the specific vaccine for safety reasons or if it is possible to continue with the recruitment of the subjects of the corresponding vaccine evaluated.

B) The randomized, double-blind, placebo-controlled phase will begin when the safety committee, after having evaluated the information of the sentinel group of the first three subjects (by vaccine and by specific route of administration), gives the authorization to continue with the recruitment. From that moment on, the subjects with the corresponding vaccination history will be randomized to receive placebo or the AVX/COVID-12 vaccine in either of the two administration arms (intramuscular or intranasal) in such a way that the total number of subjects recruited of the study for this vaccine are distributed as close as possible to 1:1 vaccine: placebo, and in equilibrium between the intramuscular and intranasal arms.

C) Specific recruitment considerations (see also sample size calculation below): To allow exploratory analyzes to be carried out for each route to be tested, by vaccine technology group or by vaccine, guiding objectives (not absolute) will be for the recruitment of 66 subjects with a history of vaccination with adenoviral technologies, 66 subjects with mRNA technologies and 66 subjects with inactivated virus technologies.

D) At the end of the study period necessary to meet the primary efficacy criterion of the study (14 days after administration of the AVX/COVID-12 vaccine or placebo), the subjects who received placebo will be masked. These subjects will receive an additional dose of the COVID-19 vaccine (ChAdOx-1-S[recombinant]) intramuscularly, and immune response parameters will be reassessed in the same manner as during the double-blind phase of the study. From that moment on, all follow-ups will continue as for the arm that originally received the AVX/COVID-12 vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 18 years old.
2. Indistinct sex.
3. Having given their informed consent.
4. No respiratory problems during the last 21 days prior to administration of the single dose.
5. No conditions or alterations in the physical examination, laboratory values and cabinet that in the opinion of the investigator may interfere with the participation of the subject in the study or require a more detailed medical study.
6. Negative PCR test for SARS-CoV-2 during the screening visit.
7. Negative pregnancy test in women with pregnancy potential.
8. Signature of commitment for the use of highly effective contraceptive methods for at least 30 days after administration of the intramuscular injection or intranasal.
9. In case of presenting any chronic disease with medical management, it must be controlled and stable without changes in treatment during the last three months prior to the scrutiny visit.
10. Commitment to maintain adequate prevention measures to avoid the contagion by SARS-CoV-2 during their participation in the study, considering themselves these strict use during the first 14 days after the baseline visit (Use of face masks in closed places, social distancing measures in spaces open, and frequent hand washing).
11. Present detectable titers of anti-Spike IgG in peripheral serum during the visit of screening with titers less than 1,200 U/mL in a chemiluminescence test.
12. Submit proof of vaccination 4 months or more after the last vaccination
13. Have been vaccinated with the complete program of any of the following vaccines against SARS-CoV-2:

    * ModeRNA
    * Pfizer
    * AstraZeneca
    * CanSino
    * Sinovac
    * Sinopharm
    * Johnson & Johnson (Janssen)
    * Sputnik V

Exclusion Criteria:

1. History of hypersensitivity or allergy to any of the components of the vaccine.
2. History of severe anaphylactic reactions from any cause.
3. History of seizures.
4. Uncontrolled chronic diseases.
5. Chronic diseases that require management with immunosuppressive agents or immune response modulators (eg, systemic corticosteroids, cyclosporine, rituximab among others).
6. Oncological disease.
7. Active participation, or during the last 3 months in any other clinical study or research experimental intervention.
8. Use within 30 days prior to screening evaluation of any drug or herbal supplement, or alternative medicine (for example, transfer factor, chlorine dioxide, etc.) aimed at treating or preventing complications or contagion by SARS-CoV-2, or any other condition.
9. Febrile illness at the time of the screening visit.
10. Have received any vaccine (experimental or approved) during the 60 days prior to the scrutiny visit.
11. Having received a blood transfusion or blood components during the last 4 months prior to the scrutiny hearing.
12. Have been a plasma donor during the last 4 months prior to the visit of scrutiny.
13. Have undergone dialysis or hemodialysis procedures during the last year prior to the scrutiny visit.
14. Work on poultry or gamecock farms.
15. History of substance abuse problems that in the opinion of the investigator could interfere with the subject's ability to adequately comply with the protocol guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Titers of circulating anti SARS-CoV-2 antibodies | Day 14
  Serum IgG, neutralizing antibodies
T-cell elicited responses | Day 14
  Percentage of cells expressing IL2, TNFalpha and IFNgamma by Flow cytometry after challenge with spike protein

SECONDARY OUTCOMES:
Titers of circulating anti SARS-CoV-2 antibodies | Day 0
  Serum IgG, neutralizing antibodies
Titers of circulating anti SARS-CoV-2 antibodies | Day 42
  Serum IgG, neutralizing antibodies
Titers of circulating anti SARS-CoV-2 antibodies | Day 90
  Serum IgG, neutralizing antibodies
Titers of circulating anti SARS-CoV-2 antibodies | Day 180
  Serum IgG, neutralizing antibodies
Titers of circulating anti SARS-CoV-2 antibodies | Day 365
  Serum IgG, neutralizing antibodies
T-cell elicited responses | Day 0
  Percentage of cells expressing IL2, TNFalpha and IFNgamma by Flow cytometry after challenge with spike protein
T-cell elicited responses | Day 180
  Percentage of cells expressing IL2, TNFalpha and IFNgamma by Flow cytometry after challenge with spike protein
T-cell elicited responses | Day 365
  Percentage of cells expressing IL2, TNFalpha and IFNgamma by Flow cytometry after challenge with spike protein

OTHER OUTCOMES:
Safety: adverse events | Day 1
  Incidence of adverse events
Safety: adverse events | Day 2
  Incidence of adverse events
Safety: adverse events | Day 3
  Incidence of adverse events
Safety: adverse events | Day 4
  Incidence of adverse events
Safety: adverse events | Day 5
  Incidence of adverse events
Safety: adverse events | Day 6
  Incidence of adverse events
Safety: adverse events | Day 7
  Incidence of adverse events
Safety: adverse events | Day 14
  Incidence of adverse events
Safety: adverse events | Day 21
  Incidence of adverse events
Safety: adverse events | Day 28
  Incidence of adverse events
Safety: adverse events | Day 42
  Incidence of adverse events
Safety: adverse events | Day 90
  Incidence of adverse events
Safety: adverse events | Day 180
  Incidence of adverse events
Safety: adverse events | Day 365
  Incidence of adverse events
Titers of circulating anti SARS-CoV-2 antibodies, Titers of circulating anti SARS-CoV-2 antibodies (IgG and neutralizing), T-cell elicited responses | Day 14
  According with to two schemes stratification as long as the number of subjects recruited allows it:
  A) By underlying technology of the vaccines received prior to the study enrollment. The three groups of technology to be explored are viruses inactivated, adenoviral vectors and technology based on mRNA. B) By specific vaccine received prior to enrollment in the study as long as the number of subjects recruited for each vaccine allows it.
Titers of mucosal IgA | Day 14
  Mucosal IgA
Titers of mucosal IgA | Day 28
  Mucosal IgA
Anti-N and anti-S antibodies | Day -4
  Appearance of anti-N and anti-S antibodies
Anti-N and anti-S antibodies | Day 7
  Appearance of anti-N and anti-S antibodies
Anti-N and anti-S antibodies | Day 14
  Appearance of anti-N and anti-S antibodies
Anti-N and anti-S antibodies | Day 42
  Appearance of anti-N and anti-S antibodies
Anti-N and anti-S antibodies | Day 90
  Appearance of anti-N and anti-S antibodies
Anti-N and anti-S antibodies | Day 180
  Appearance of anti-N and anti-S antibodies
Anti-N and anti-S antibodies | Day 365
  Appearance of anti-N and anti-S antibodies
Incidence of confirmed cases of SARS-CoV-2 infection | Day 28 until the end of the study
  Evaluation of the incidence of confirmed cases of SARS-CoV-2 infection in study subjects from systematic vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Laura Castro, MD, Principal Investigator — CAIMED Investigación en Salud S.A. de C.V.; Niels Hansen, MD, Principal Investigator — Unidad Médico Familiar No. 20 Instituto Mexicano del Seguro Social
Locations (4):
- Mexico (4):
  - Centro Mexicano de Estudios Clínicos CEMDEC SA de CV, Mexico City, Mexico City
  - CAIMED Investigación en Salud S.A. de C.V., Mexico City, Mexico City
  - Unidad Médico Familiar No. 20 Instituto Mexicano del Seguro Social, Mexico City, Mexico City
  - Oaxaca Site Management Organization S.C., Oaxaca City, Oaxaca

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data (including data dictionaries) will not be shared, but only to the extent permitted in the informed consent and under Mexican law.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available immediately following publication and for 12 months thereafter.
Access Criteria: Data will be available only to investigators whose proposed use of the data has been authorized by an independent review committee and the ethics committees involved in the authorization of the protocol, and/or the Federal Commission for the Protection against Sanitary Risks (COFEPRIS) in Mexico if required by law. The permitted use of the data will be as authorized. Proposals or requests should be directed to gustavo.peralta@avimex.com.mx and authorized data requestors must sign a data access agreement.

REFERENCES:
- [Background] Logunov DY, Dolzhikova IV, Zubkova OV, Tukhvatullin AI, Shcheblyakov DV, Dzharullaeva AS, Grousova DM, Erokhova AS, Kovyrshina AV, Botikov AG, Izhaeva FM, Popova O, Ozharovskaya TA, Esmagambetov IB, Favorskaya IA, Zrelkin DI, Voronina DV, Shcherbinin DN, Semikhin AS, Simakova YV, Tokarskaya EA, Lubenets NL, Egorova DA, Shmarov MM, Nikitenko NA, Morozova LF, Smolyarchuk EA, Kryukov EV, Babira VF, Borisevich SV, Naroditsky BS, Gintsburg AL. Safety and immunogenicity of an rAd26 and rAd5 vector-based heterologous prime-boost COVID-19 vaccine in two formulations: two open, non-randomised phase 1/2 studies from Russia. Lancet. 2020 Sep 26;396(10255):887-897. doi: 10.1016/S0140-6736(20)31866-3. Epub 2020 Sep 4. PMID 32896291
- [Background] Dhillon P, Altmann D, Male V. COVID-19 vaccines: what do we know so far? FEBS J. 2021 Sep;288(17):4996-5009. doi: 10.1111/febs.16094. Epub 2021 Jul 19. PMID 34288409
- [Background] Zamai L, Rocchi MBL. Hypothesis: Possible influence of antivector immunity and SARS-CoV-2 variants on efficacy of ChAdOx1 nCoV-19 vaccine. Br J Pharmacol. 2022 Jan;179(2):218-226. doi: 10.1111/bph.15620. Epub 2021 Jul 31. PMID 34331459
- [Background] Barros-Martins J, Hammerschmidt SI, Cossmann A, Odak I, Stankov MV, Morillas Ramos G, Dopfer-Jablonka A, Heidemann A, Ritter C, Friedrichsen M, Schultze-Florey C, Ravens I, Willenzon S, Bubke A, Ristenpart J, Janssen A, Ssebyatika G, Bernhardt G, Munch J, Hoffmann M, Pohlmann S, Krey T, Bosnjak B, Forster R, Behrens GMN. Immune responses against SARS-CoV-2 variants after heterologous and homologous ChAdOx1 nCoV-19/BNT162b2 vaccination. Nat Med. 2021 Sep;27(9):1525-1529. doi: 10.1038/s41591-021-01449-9. Epub 2021 Jul 14. PMID 34262158
- [Background] He Q, Mao Q, An C, Zhang J, Gao F, Bian L, Li C, Liang Z, Xu M, Wang J. Heterologous prime-boost: breaking the protective immune response bottleneck of COVID-19 vaccine candidates. Emerg Microbes Infect. 2021 Dec;10(1):629-637. doi: 10.1080/22221751.2021.1902245. PMID 33691606
- [Background] Normark J, Vikstrom L, Gwon YD, Persson IL, Edin A, Bjorsell T, Dernstedt A, Christ W, Tevell S, Evander M, Klingstrom J, Ahlm C, Forsell M. Heterologous ChAdOx1 nCoV-19 and mRNA-1273 Vaccination. N Engl J Med. 2021 Sep 9;385(11):1049-1051. doi: 10.1056/NEJMc2110716. Epub 2021 Jul 14. No abstract available. PMID 34260850
- [Background] Hill JA, Ujjani CS, Greninger AL, Shadman M, Gopal AK. Immunogenicity of a heterologous COVID-19 vaccine after failed vaccination in a lymphoma patient. Cancer Cell. 2021 Aug 9;39(8):1037-1038. doi: 10.1016/j.ccell.2021.06.015. Epub 2021 Jun 26. No abstract available. PMID 34242571
- [Background] Velasco M, Galan MI, Casas ML, Perez-Fernandez E, Martinez-Ponce D, Gonzalez-Pineiro B, Castilla V, Guijarro C; Alcorcon COVID-19 Working Group. Impact of Previous Coronavirus Disease 2019 on Immune Response After a Single Dose of BNT162b2 Severe Acute Respiratory Syndrome Coronavirus 2 Vaccine. Open Forum Infect Dis. 2021 Jun 4;8(7):ofab299. doi: 10.1093/ofid/ofab299. eCollection 2021 Jul. PMID 34258322
- [Background] Levi R, Azzolini E, Pozzi C, Ubaldi L, Lagioia M, Mantovani A, Rescigno M. One dose of SARS-CoV-2 vaccine exponentially increases antibodies in individuals who have recovered from symptomatic COVID-19. J Clin Invest. 2021 Jun 15;131(12):e149154. doi: 10.1172/JCI149154. PMID 33956667
- [Background] Reynolds CJ, Pade C, Gibbons JM, Butler DK, Otter AD, Menacho K, Fontana M, Smit A, Sackville-West JE, Cutino-Moguel T, Maini MK, Chain B, Noursadeghi M; UK COVIDsortium Immune Correlates Network; Brooks T, Semper A, Manisty C, Treibel TA, Moon JC; UK COVIDsortium Investigators; Valdes AM, McKnight A, Altmann DM, Boyton R. Prior SARS-CoV-2 infection rescues B and T cell responses to variants after first vaccine dose. Science. 2021 Apr 30;372(6549):1418-23. doi: 10.1126/science.abh1282. Online ahead of print. PMID 33931567
- [Background] Sun W, Leist SR, McCroskery S, Liu Y, Slamanig S, Oliva J, Amanat F, Schafer A, Dinnon KH 3rd, Garcia-Sastre A, Krammer F, Baric RS, Palese P. Newcastle disease virus (NDV) expressing the spike protein of SARS-CoV-2 as a live virus vaccine candidate. EBioMedicine. 2020 Dec;62:103132. doi: 10.1016/j.ebiom.2020.103132. Epub 2020 Nov 21. PMID 33232870
- [Background] DiNapoli JM, Kotelkin A, Yang L, Elankumaran S, Murphy BR, Samal SK, Collins PL, Bukreyev A. Newcastle disease virus, a host range-restricted virus, as a vaccine vector for intranasal immunization against emerging pathogens. Proc Natl Acad Sci U S A. 2007 Jun 5;104(23):9788-93. doi: 10.1073/pnas.0703584104. Epub 2007 May 29. PMID 17535926
- [Background] Bukreyev A, Huang Z, Yang L, Elankumaran S, St Claire M, Murphy BR, Samal SK, Collins PL. Recombinant newcastle disease virus expressing a foreign viral antigen is attenuated and highly immunogenic in primates. J Virol. 2005 Nov;79(21):13275-84. doi: 10.1128/JVI.79.21.13275-13284.2005. PMID 16227250
- [Background] Brown CM, Vostok J, Johnson H, Burns M, Gharpure R, Sami S, Sabo RT, Hall N, Foreman A, Schubert PL, Gallagher GR, Fink T, Madoff LC, Gabriel SB, MacInnis B, Park DJ, Siddle KJ, Harik V, Arvidson D, Brock-Fisher T, Dunn M, Kearns A, Laney AS. Outbreak of SARS-CoV-2 Infections, Including COVID-19 Vaccine Breakthrough Infections, Associated with Large Public Gatherings - Barnstable County, Massachusetts, July 2021. MMWR Morb Mortal Wkly Rep. 2021 Aug 6;70(31):1059-1062. doi: 10.15585/mmwr.mm7031e2. PMID 34351882
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Chan JF, Yuan S, Kok KH, To KK, Chu H, Yang J, Xing F, Liu J, Yip CC, Poon RW, Tsoi HW, Lo SK, Chan KH, Poon VK, Chan WM, Ip JD, Cai JP, Cheng VC, Chen H, Hui CK, Yuen KY. A familial cluster of pneumonia associated with the 2019 novel coronavirus indicating person-to-person transmission: a study of a family cluster. Lancet. 2020 Feb 15;395(10223):514-523. doi: 10.1016/S0140-6736(20)30154-9. Epub 2020 Jan 24. PMID 31986261
- [Background] Chan JF, Kok KH, Zhu Z, Chu H, To KK, Yuan S, Yuen KY. Genomic characterization of the 2019 novel human-pathogenic coronavirus isolated from a patient with atypical pneumonia after visiting Wuhan. Emerg Microbes Infect. 2020 Jan 28;9(1):221-236. doi: 10.1080/22221751.2020.1719902. eCollection 2020. PMID 31987001
- [Background] Wu F, Zhao S, Yu B, Chen YM, Wang W, Song ZG, Hu Y, Tao ZW, Tian JH, Pei YY, Yuan ML, Zhang YL, Dai FH, Liu Y, Wang QM, Zheng JJ, Xu L, Holmes EC, Zhang YZ. A new coronavirus associated with human respiratory disease in China. Nature. 2020 Mar;579(7798):265-269. doi: 10.1038/s41586-020-2008-3. Epub 2020 Feb 3. PMID 32015508
- [Background] Wan Y, Shang J, Graham R, Baric RS, Li F. Receptor Recognition by the Novel Coronavirus from Wuhan: an Analysis Based on Decade-Long Structural Studies of SARS Coronavirus. J Virol. 2020 Mar 17;94(7):e00127-20. doi: 10.1128/JVI.00127-20. Print 2020 Mar 17. PMID 31996437
- [Background] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651
- [Background] Yao H, Song Y, Chen Y, Wu N, Xu J, Sun C, Zhang J, Weng T, Zhang Z, Wu Z, Cheng L, Shi D, Lu X, Lei J, Crispin M, Shi Y, Li L, Li S. Molecular Architecture of the SARS-CoV-2 Virus. Cell. 2020 Oct 29;183(3):730-738.e13. doi: 10.1016/j.cell.2020.09.018. Epub 2020 Sep 6. PMID 32979942
- [Background] Wrapp D, Wang N, Corbett KS, Goldsmith JA, Hsieh CL, Abiona O, Graham BS, McLellan JS. Cryo-EM structure of the 2019-nCoV spike in the prefusion conformation. Science. 2020 Mar 13;367(6483):1260-1263. doi: 10.1126/science.abb2507. Epub 2020 Feb 19. PMID 32075877
- [Background] Piccoli L, Park YJ, Tortorici MA, Czudnochowski N, Walls AC, Beltramello M, Silacci-Fregni C, Pinto D, Rosen LE, Bowen JE, Acton OJ, Jaconi S, Guarino B, Minola A, Zatta F, Sprugasci N, Bassi J, Peter A, De Marco A, Nix JC, Mele F, Jovic S, Rodriguez BF, Gupta SV, Jin F, Piumatti G, Lo Presti G, Pellanda AF, Biggiogero M, Tarkowski M, Pizzuto MS, Cameroni E, Havenar-Daughton C, Smithey M, Hong D, Lepori V, Albanese E, Ceschi A, Bernasconi E, Elzi L, Ferrari P, Garzoni C, Riva A, Snell G, Sallusto F, Fink K, Virgin HW, Lanzavecchia A, Corti D, Veesler D. Mapping Neutralizing and Immunodominant Sites on the SARS-CoV-2 Spike Receptor-Binding Domain by Structure-Guided High-Resolution Serology. Cell. 2020 Nov 12;183(4):1024-1042.e21. doi: 10.1016/j.cell.2020.09.037. Epub 2020 Sep 16. PMID 32991844
- [Background] Tan CW, Chia WN, Qin X, Liu P, Chen MI, Tiu C, Hu Z, Chen VC, Young BE, Sia WR, Tan YJ, Foo R, Yi Y, Lye DC, Anderson DE, Wang LF. A SARS-CoV-2 surrogate virus neutralization test based on antibody-mediated blockage of ACE2-spike protein-protein interaction. Nat Biotechnol. 2020 Sep;38(9):1073-1078. doi: 10.1038/s41587-020-0631-z. Epub 2020 Jul 23. PMID 32704169
- [Background] Chen X, Pan Z, Yue S, Yu F, Zhang J, Yang Y, Li R, Liu B, Yang X, Gao L, Li Z, Lin Y, Huang Q, Xu L, Tang J, Hu L, Zhao J, Liu P, Zhang G, Chen Y, Deng K, Ye L. Disease severity dictates SARS-CoV-2-specific neutralizing antibody responses in COVID-19. Signal Transduct Target Ther. 2020 Sep 2;5(1):180. doi: 10.1038/s41392-020-00301-9. PMID 32879307
- [Background] Liu L, To KK, Chan KH, Wong YC, Zhou R, Kwan KY, Fong CH, Chen LL, Choi CY, Lu L, Tsang OT, Leung WS, To WK, Hung IF, Yuen KY, Chen Z. High neutralizing antibody titer in intensive care unit patients with COVID-19. Emerg Microbes Infect. 2020 Dec;9(1):1664-1670. doi: 10.1080/22221751.2020.1791738. PMID 32618497
- [Background] Choe PG, Kang CK, Suh HJ, Jung J, Kang E, Lee SY, Song KH, Kim HB, Kim NJ, Park WB, Kim ES, Oh MD. Antibody Responses to SARS-CoV-2 at 8 Weeks Postinfection in Asymptomatic Patients. Emerg Infect Dis. 2020 Oct;26(10):2484-2487. doi: 10.3201/eid2610.202211. Epub 2020 Jun 24. PMID 32579877
- [Background] Le Bert N, Tan AT, Kunasegaran K, Tham CYL, Hafezi M, Chia A, Chng MHY, Lin M, Tan N, Linster M, Chia WN, Chen MI, Wang LF, Ooi EE, Kalimuddin S, Tambyah PA, Low JG, Tan YJ, Bertoletti A. SARS-CoV-2-specific T cell immunity in cases of COVID-19 and SARS, and uninfected controls. Nature. 2020 Aug;584(7821):457-462. doi: 10.1038/s41586-020-2550-z. Epub 2020 Jul 15. PMID 32668444
- [Background] Dessie ZG, Zewotir T. Mortality-related risk factors of COVID-19: a systematic review and meta-analysis of 42 studies and 423,117 patients. BMC Infect Dis. 2021 Aug 21;21(1):855. doi: 10.1186/s12879-021-06536-3. PMID 34418980
- [Background] Wang Y, Perlman S. COVID-19: Inflammatory Profile. Annu Rev Med. 2022 Jan 27;73:65-80. doi: 10.1146/annurev-med-042220-012417. Epub 2021 Aug 26. PMID 34437814
- [Background] Wagner C, Griesel M, Mikolajewska A, Mueller A, Nothacker M, Kley K, Metzendorf MI, Fischer AL, Kopp M, Stegemann M, Skoetz N, Fichtner F. Systemic corticosteroids for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Aug 16;8(8):CD014963. doi: 10.1002/14651858.CD014963. PMID 34396514
- [Background] Ansems K, Grundeis F, Dahms K, Mikolajewska A, Thieme V, Piechotta V, Metzendorf MI, Stegemann M, Benstoem C, Fichtner F. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD014962. doi: 10.1002/14651858.CD014962. PMID 34350582
- [Background] Ghosn L, Chaimani A, Evrenoglou T, Davidson M, Grana C, Schmucker C, Bollig C, Henschke N, Sguassero Y, Nejstgaard CH, Menon S, Nguyen TV, Ferrand G, Kapp P, Riveros C, Avila C, Devane D, Meerpohl JJ, Rada G, Hrobjartsson A, Grasselli G, Tovey D, Ravaud P, Boutron I. Interleukin-6 blocking agents for treating COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 Mar 18;3(3):CD013881. doi: 10.1002/14651858.CD013881. PMID 33734435
- [Background] Khoury DS, Cromer D, Reynaldi A, Schlub TE, Wheatley AK, Juno JA, Subbarao K, Kent SJ, Triccas JA, Davenport MP. Neutralizing antibody levels are highly predictive of immune protection from symptomatic SARS-CoV-2 infection. Nat Med. 2021 Jul;27(7):1205-1211. doi: 10.1038/s41591-021-01377-8. Epub 2021 May 17. PMID 34002089
- [Background] Liu A, Li Y, Peng J, Huang Y, Xu D. Antibody responses against SARS-CoV-2 in COVID-19 patients. J Med Virol. 2021 Jan;93(1):144-148. doi: 10.1002/jmv.26241. Epub 2020 Aug 2. No abstract available. PMID 32603501
- [Background] Perreault J, Tremblay T, Fournier MJ, Drouin M, Beaudoin-Bussieres G, Prevost J, Lewin A, Begin P, Finzi A, Bazin R. Waning of SARS-CoV-2 RBD antibodies in longitudinal convalescent plasma samples within 4 months after symptom onset. Blood. 2020 Nov 26;136(22):2588-2591. doi: 10.1182/blood.2020008367. PMID 33001206
- [Background] Post N, Eddy D, Huntley C, van Schalkwyk MCI, Shrotri M, Leeman D, Rigby S, Williams SV, Bermingham WH, Kellam P, Maher J, Shields AM, Amirthalingam G, Peacock SJ, Ismail SA. Antibody response to SARS-CoV-2 infection in humans: A systematic review. PLoS One. 2020 Dec 31;15(12):e0244126. doi: 10.1371/journal.pone.0244126. eCollection 2020. PMID 33382764
- [Background] Juthani PV, Gupta A, Borges KA, Price CC, Lee AI, Won CH, Chun HJ. Hospitalisation among vaccine breakthrough COVID-19 infections. Lancet Infect Dis. 2021 Nov;21(11):1485-1486. doi: 10.1016/S1473-3099(21)00558-2. Epub 2021 Sep 7. No abstract available. PMID 34506735
- [Background] Patalon T, Gazit S, Pitzer VE, Prunas O, Warren JL, Weinberger DM. Odds of Testing Positive for SARS-CoV-2 Following Receipt of 3 vs 2 Doses of the BNT162b2 mRNA Vaccine. JAMA Intern Med. 2022 Feb 1;182(2):179-184. doi: 10.1001/jamainternmed.2021.7382. PMID 34846533
- [Background] Borobia AM, Carcas AJ, Perez-Olmeda M, Castano L, Bertran MJ, Garcia-Perez J, Campins M, Portoles A, Gonzalez-Perez M, Garcia Morales MT, Arana-Arri E, Aldea M, Diez-Fuertes F, Fuentes I, Ascaso A, Lora D, Imaz-Ayo N, Baron-Mira LE, Agusti A, Perez-Ingidua C, Gomez de la Camara A, Arribas JR, Ochando J, Alcami J, Belda-Iniesta C, Frias J; CombiVacS Study Group. Immunogenicity and reactogenicity of BNT162b2 booster in ChAdOx1-S-primed participants (CombiVacS): a multicentre, open-label, randomised, controlled, phase 2 trial. Lancet. 2021 Jul 10;398(10295):121-130. doi: 10.1016/S0140-6736(21)01420-3. Epub 2021 Jun 25. PMID 34181880
- [Background] Hsieh CL, Goldsmith JA, Schaub JM, DiVenere AM, Kuo HC, Javanmardi K, Le KC, Wrapp D, Lee AG, Liu Y, Chou CW, Byrne PO, Hjorth CK, Johnson NV, Ludes-Meyers J, Nguyen AW, Park J, Wang N, Amengor D, Lavinder JJ, Ippolito GC, Maynard JA, Finkelstein IJ, McLellan JS. Structure-based design of prefusion-stabilized SARS-CoV-2 spikes. Science. 2020 Sep 18;369(6510):1501-1505. doi: 10.1126/science.abd0826. Epub 2020 Jul 23. PMID 32703906
- [Background] Rodda LB, Netland J, Shehata L, Pruner KB, Morawski PA, Thouvenel CD, Takehara KK, Eggenberger J, Hemann EA, Waterman HR, Fahning ML, Chen Y, Hale M, Rathe J, Stokes C, Wrenn S, Fiala B, Carter L, Hamerman JA, King NP, Gale M Jr, Campbell DJ, Rawlings DJ, Pepper M. Functional SARS-CoV-2-Specific Immune Memory Persists after Mild COVID-19. Cell. 2021 Jan 7;184(1):169-183.e17. doi: 10.1016/j.cell.2020.11.029. Epub 2020 Nov 23. PMID 33296701
- [Background] Barouch DH, Stephenson KE, Sadoff J, Yu J, Chang A, Gebre M, McMahan K, Liu J, Chandrashekar A, Patel S, Le Gars M, de Groot AM, Heerwegh D, Struyf F, Douoguih M, van Hoof J, Schuitemaker H. Durable Humoral and Cellular Immune Responses 8 Months after Ad26.COV2.S Vaccination. N Engl J Med. 2021 Sep 2;385(10):951-953. doi: 10.1056/NEJMc2108829. Epub 2021 Jul 14. No abstract available. PMID 34260834
- [Background] Thomas SJ, Moreira ED Jr, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Polack FP, Zerbini C, Bailey R, Swanson KA, Xu X, Roychoudhury S, Koury K, Bouguermouh S, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Yang Q, Liberator P, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Gruber WC, Jansen KU; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine through 6 Months. N Engl J Med. 2021 Nov 4;385(19):1761-1773. doi: 10.1056/NEJMoa2110345. Epub 2021 Sep 15. PMID 34525277
- [Background] Lopez Bernal J, Andrews N, Gower C, Gallagher E, Simmons R, Thelwall S, Stowe J, Tessier E, Groves N, Dabrera G, Myers R, Campbell CNJ, Amirthalingam G, Edmunds M, Zambon M, Brown KE, Hopkins S, Chand M, Ramsay M. Effectiveness of Covid-19 Vaccines against the B.1.617.2 (Delta) Variant. N Engl J Med. 2021 Aug 12;385(7):585-594. doi: 10.1056/NEJMoa2108891. Epub 2021 Jul 21. PMID 34289274
- [Background] Hacisuleyman E, Hale C, Saito Y, Blachere NE, Bergh M, Conlon EG, Schaefer-Babajew DJ, DaSilva J, Muecksch F, Gaebler C, Lifton R, Nussenzweig MC, Hatziioannou T, Bieniasz PD, Darnell RB. Vaccine Breakthrough Infections with SARS-CoV-2 Variants. N Engl J Med. 2021 Jun 10;384(23):2212-2218. doi: 10.1056/NEJMoa2105000. Epub 2021 Apr 21. PMID 33882219
- [Background] Bergwerk M, Gonen T, Lustig Y, Amit S, Lipsitch M, Cohen C, Mandelboim M, Levin EG, Rubin C, Indenbaum V, Tal I, Zavitan M, Zuckerman N, Bar-Chaim A, Kreiss Y, Regev-Yochay G. Covid-19 Breakthrough Infections in Vaccinated Health Care Workers. N Engl J Med. 2021 Oct 14;385(16):1474-1484. doi: 10.1056/NEJMoa2109072. Epub 2021 Jul 28. PMID 34320281
- [Background] Keehner J, Horton LE, Binkin NJ, Laurent LC; SEARCH Alliance; Pride D, Longhurst CA, Abeles SR, Torriani FJ. Resurgence of SARS-CoV-2 Infection in a Highly Vaccinated Health System Workforce. N Engl J Med. 2021 Sep 30;385(14):1330-1332. doi: 10.1056/NEJMc2112981. Epub 2021 Sep 1. No abstract available. PMID 34469645
- [Background] Mathieu E, Ritchie H, Ortiz-Ospina E, Roser M, Hasell J, Appel C, Giattino C, Rodes-Guirao L. A global database of COVID-19 vaccinations. Nat Hum Behav. 2021 Jul;5(7):947-953. doi: 10.1038/s41562-021-01122-8. Epub 2021 May 10. PMID 33972767
- [Background] Macpherson LW. Some Observations On The Epizootiology Of NewCastle Disease. Can J Comp Med Vet Sci. 1956 May;20(5):155-68. No abstract available. PMID 17648892
- [Background] Alexander DJ. Newcastle disease and other avian paramyxoviruses. Rev Sci Tech. 2000 Aug;19(2):443-62. doi: 10.20506/rst.19.2.1231. PMID 10935273
- [Background] NELSON CB, POMEROY BS, SCHRALL K, PARK WE, LINDEMAN RJ. An outbreak of conjunctivitis due to Newcastle disease virus (NDV) occurring in poultry workers. Am J Public Health Nations Health. 1952 Jun;42(6):672-8. doi: 10.2105/ajph.42.6.672. No abstract available. PMID 14924001
- [Background] Kim SH, Samal SK. Newcastle Disease Virus as a Vaccine Vector for Development of Human and Veterinary Vaccines. Viruses. 2016 Jul 4;8(7):183. doi: 10.3390/v8070183. PMID 27384578
- [Background] Sun W, McCroskery S, Liu WC, Leist SR, Liu Y, Albrecht RA, Slamanig S, Oliva J, Amanat F, Schafer A, Dinnon KH 3rd, Innis BL, Garcia-Sastre A, Krammer F, Baric RS, Palese P. A Newcastle Disease Virus (NDV) Expressing a Membrane-Anchored Spike as a Cost-Effective Inactivated SARS-CoV-2 Vaccine. Vaccines (Basel). 2020 Dec 17;8(4):771. doi: 10.3390/vaccines8040771. PMID 33348607
- [Background] Naranjo CA, Busto U, Sellers EM, Sandor P, Ruiz I, Roberts EA, Janecek E, Domecq C, Greenblatt DJ. A method for estimating the probability of adverse drug reactions. Clin Pharmacol Ther. 1981 Aug;30(2):239-45. doi: 10.1038/clpt.1981.154. No abstract available. PMID 7249508
- [Derived] Lopez-Macias C, Torres M, Armenta-Copca B, Wacher NH, Castro-Castrezana L, Colli-Dominguez AA, Rivera-Hernandez T, Torres-Flores A, Damian-Hernandez M, Ramirez-Martinez L, la Rosa GP, Rojas-Martinez O, Suarez-Martinez A, Peralta-Sanchez G, Carranza C, Juarez E, Zamudio-Meza H, Carreto-Binaghi LE, Viettri M, Romero-Rodriguez D, Palencia A, Reyna-Rosas E, Marquez-Garcia JE, Sarfati-Mizrahi D, Sun W, Chagoya-Cortes HE, Castro-Peralta F, Palese P, Krammer F, Garcia-Sastre A, Lozano-Dubernard B. Phase II study on the safety and immunogenicity of single-dose intramuscular or intranasal administration of the AVX/COVID-12 "Patria" recombinant Newcastle disease virus vaccine as a heterologous booster against COVID-19 in Mexico. Vaccine. 2025 Jan 1;43(Pt 2):126511. doi: 10.1016/j.vaccine.2024.126511. Epub 2024 Nov 10. PMID 39527880
- [Derived] Nakahashi-Ouchida R, Fujihashi K, Kurashima Y, Yuki Y, Kiyono H. Nasal vaccines: solutions for respiratory infectious diseases. Trends Mol Med. 2023 Feb;29(2):124-140. doi: 10.1016/j.molmed.2022.10.009. Epub 2022 Nov 23. PMID 36435633